CLINICAL TRIAL: NCT02266511
Title: A Single-dose, Randomized, Two-treatment, Two-period, Open-label, Crossover Study to Assess the Bioequivalence of Two Batches of Tamsulosin Hydrochloride 0.4-mg Capsules in Healthy Male Subjects
Brief Title: Study to Assess the Bioequivalence of Two Batches of Tamsulosin Hydrochloride in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 527.22
Record Dates: First submitted 2014-10-16; First posted 2014-10-17 (Estimated); Last update posted 2014-10-17 (Estimated); Status verified 2014-10

CONDITIONS: Healthy
MeSH Terms: interventions — Tamsulosin

ARMS (2):
- Sequence 1 (Experimental): Flomax®, Nishine facility followed by Flomax®, Norman II facility
  Interventions: Drug: Flomax®, Norman II facility; Drug: Flomax®, Nishine facility
- Sequence 2 (Experimental): Flomax®, Norman II facility followed by Flomax®, Nishine facility
  Interventions: Drug: Flomax®, Norman II facility; Drug: Flomax®, Nishine facility

INTERVENTIONS:
Drug: Flomax®, Norman II facility
  Other Names: Tamsulosin hydrochloride
Drug: Flomax®, Nishine facility
  Other Names: Tamsulosin hydrochloride

SUMMARY:
The objective of this study is to determine the bioequivalence of two batches of Flomax® 0.4 mg capsules in healthy male subjects. One is a commercial scale batch produced at the Nishine facility, and the other is a batch, of equal size, produced at the Norman II facility

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consents, as evidenced by signature on an Informed Consent Form approved by the investigational review board (IRB) following a full explanation of the nature and purpose of the study
* Be a healthy male of any race between 18 and 40 years of age
* Have a body weight within 10 % of normal for sex, height, and frame as specified by the Body Weight Nomogram for Inclusion/Exclusion Criteria
* Have no clinically significant abnormalities o the basis of medical history, physical examination, and vital signs with no significant orthostatic blood pressure change, which is defined as no more than a 20 mm Hg drop in systolic blood pressure on assuming and maintaining the standing position for 3 minutes after being supine for at least 5 minutes. There should be no clinically significant symptoms associated with the orthostatic blood pressure testing procedure
* Have cardiovascular system that is within normal limits based on history, physical examination, and a 12-lead electrocardiogram (ECG)
* Have a negative test for ethanol by breathalyzer
* Have the ability to understand the requirements of the study, agree to abide by the study restrictions, and agree to return for the required assessments

Exclusion Criteria:

* Require ambulatory assistance (e.g., canes or walkers)
* Have a history of a "first dose hypotensive episode" upon starting therapy with an alpha-blocker
* Have a history of a pathological fall (unintentional change in body position) during the last year occurring under circumstances in which normal homeostatic mechanisms would ordinarily maintain stability or syncope
* Have any medical or laboratory abnormalities (liver function tests, blood urea nitrogen, and creatinine should not be outside the reference range for the clinical laboratory). Any subject who enters into the study with laboratory abnormalities must be approved by the Medical Monitor prior to enrollment
* Have abnormal alpha-1-acid glycoprotein values (i.e., values greater than 120 mg/dL)
* Have any history of acute angina attacks during the prior 6 months
* Have any abnormality of the ECG or a history of a documented myocardial infarction (electrocardiographic changes, serum enzymes increases, and hospitalization) during the prior 6 months, or evidence of any myocardial infarction on an ECG
* Have a New York Heart Association's Functional Classification of Heart Failure Class I, II, III, or IV
* Have a prior history of endocarditis
* Use any prescription medications within 2 weeks of dosing, or over-the-counter concomitant therapies with the exception of vitamins, dietary supplements, and acetaminophen within 7 days of dosing
* Have used an investigational drug within 1 month (30 days) of the Screening Period visit
* Donated blood within 1 month of entering study
* Have a known history of any of the following:

  * Clinically significant renal disease (renal dysfunction; i.e., creatinine greater than or equal to 2.0 mg/dL)
  * Severe cardiovascular disease (coarctation of the aorta, severe cardiac failure, second or third degree heart block, or severe angina)
  * Pulmonary disease (chronic lung disease or emphysema of a degree that could cause functional abnormalities of the right heart)
* Have acute illness (e.g., acute upper respiratory infection) within 2 weeks prior to the start of the study
* Have any medical condition that might interfere with either the absorption, distribution, metabolism, or excretion of tamsulosin
* Have a history of any illness or allergy that, in the opinion of the Investigator, might confound the results of the study or pose additional risk in administering Flomax® to the subject
* Have a history of liver disease or any physical findings suggestive of liver disease
* Have smoked within the last 3 months or be known as or be suspected as an alcohol abuser or illicit drug user within the past year, or have a positive urine drug screen
* Exhibit, in the opinion of the Investigator, the signs or symptoms of an immunodeficiency syndrome, whether spontaneously acquired, congenital, or iatrogenic (These syndromes are characterized by unusual susceptibility to infection [bacterial, viral, or fungal], the occurrence of autoimmune disease, and lymphoreticular malignancies)
* Have calculated creatinine clearance less than 90 mL/min based upon the following formula:

  * Creatinine Clearance = (140 - age in years) (weight in kg) / (72) (serum creatinine)
* Have a history of cancer except for nonmelanoma skin cancer treated by excision

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 1999-08; Primary Completion 1999-09 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve of the analyte in plasma at different time points (AUC) | Up to 48 h after drug administration
Maximum concentration of the analyte in plasma (Cmax) | Up to 48 h after drug administration
Time to reach the maximum concentration of the analyte in plasma (tmax) | Up to 48 h after drug administration
Elimination half-life (t1/2) | Up to 48 h after drug administration
Terminal elimination rate constant of the analyte in plasma (λz) | Up to 48 h after drug administration
Number of participants with clinically relevant changes in laboratory values | Up to day 3 after last drug administration
Number of participants with clinically relevant changes in vital signs (heart rate, orthostatic blood pressure, weight, temperature, respiration rate) | Up to day 3 after last drug administration
Number of participants with adverse events | Up to day 3 after last drug administration
Number of participants with clinically relevant changes in ECG | Up to day 3 after last drug administration